CLINICAL TRIAL: NCT04912947
Title: EValuation of the Antioxidant and Anti-inflammatory Capacity of Nutraceutical IMMU·SYSTEM Food Supplement (EVAANIS)
Acronym: EVAANIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Complife Italia Srl (Industry)
Collaborators: Macrofarm Srl (Industry); Icim International Srl (Unknown)
Responsible Party: Principal Investigator, FRANCESCO PUOCI, Associate Professor - DFSSN, University of Calabria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EVAANIS
Record Dates: First submitted 2021-04-28; First posted 2021-06-03 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Oxidative Stress
Keywords: Oxidative Stress; Glutathione; Immune system activity; Food supplement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Active Comparator): One cp/day of the IMMUSYSTEM food supplement for 3 months
  Interventions: Dietary Supplement: Immusystem
- Placebo (Placebo Comparator): One cp/day of Placebo for 3 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Immusystem — Dietary supplement containing: Piceid, Glycine, Glutamine, Acetylcysteine, Zinc and Vitamin B6
  Arms: Dietary supplement
Other: Placebo — Maltodextrin placebo capsule
  Arms: Placebo

SUMMARY:
The aim of the study is to verify the effectiveness of Nutraceutical IMMU·SYSTEM Dietary supplement in reducing the levels of oxidative stress and inflammation in a sample of healthy adult subjects with high baseline levels of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity;
* Age between 30 and 65 years;
* Smokers who have smoked at least 100 cigarettes in their lifetime and smoke at least 10 cigarettes a day;
* Sportsmen who have been playing sports for at least 6 months between 4 and 8 hours per week;
* Signature of informed consent.

Exclusion Criteria:

* Systemic pathologies;
* Active drug therapy;
* Estrogen-progestogen therapy;
* Pregnancy;
* Allergies to the components of the raw material under study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Erythrocytes GSH/GSSG ratio | Month 3
  Change from Baseline reduced/oxidized glutathione ratio in erythrocytes at 3 Months
Change in Erythrocytes GSH/GSSG ratio | Month 1
  Change from Baseline reduced/oxidized glutathione ratio in erythrocytes at 1st Month

SECONDARY OUTCOMES:
Change in Immune system activity | Month 3
  Change from Baseline of Serum levels of immune system activity: TNFα, IL-6, IL-2 at 3 Months
Change in Immune system activity | Month 1
  Change from Baseline of Serum levels of immune system activity: TNFα, IL-6, IL-2 at 1st Month
Change in Immune system activity | Month 3
  Change from Baseline of Serum levels of IFN-γ at 1st Month
Change in Immune system activity | Month 1
  Change from Baseline of Serum levels of IFN-γ at 1st Month

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Puoci, PhD, Principal Investigator — DFSSN - UNICAL
Locations (1):
- University of Calabria, Rende, CS, Italy